CLINICAL TRIAL: NCT05393076
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Pharmacokinetics and Safety of Linerixibat in Adults With Moderate Hepatic Impairment and Healthy Matched Control Participants
Brief Title: Phase I Study of Linerixibat in Adults With Moderate Hepatic Impairment and Healthy Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 214899
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Pruritus
Keywords: Linerixibat; Pruritus; GSK2330672; Pharmacokinetics; Primary biliary cholangitis; Hepatic impairment; Liver Cirrhosis
MeSH Terms: conditions — Pruritus; Liver Cirrhosis, Biliary; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: This phase 1 study is an open-label, non-randomized, single-dose linerixibat study with 2 cohorts (moderate hepatic impairment and matched healthy control participants).
Masking Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Moderate hepatic impairment participants) (Experimental): Eligible participants to receive single dose of linerixibat.
  Interventions: Drug: Linerixibat
- Cohort 2 (Matched healthy control participants) (Experimental): Eligible participants to receive single dose of linerixibat
  Interventions: Drug: Linerixibat

INTERVENTIONS:
Drug: Linerixibat — Linerixibat dose and administration as per study intervention.

SUMMARY:
This is a phase 1, open-label, single-dose study in adults with moderate hepatic impairment (defined as Child-Pugh B cirrhosis) and matched healthy control participants with normal hepatic function. All participants in both cohorts (moderate hepatic impairment and matched healthy controls) will receive a single dose of the study drug, linerixibat. The purpose of this study is to assess the effect of hepatic impairment on the pharmacokinetics (PK) and safety of linerixibat.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Age: 18 to 75 years of age (inclusive).
* Weight greater than (>) 45 kilograms (kg) and body mass index (BMI) 18.5 - 40 kg per square meter (kg/m^2) (inclusive).
* Male and female- A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies; not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow contraceptive guidance during the treatment period and until at least 4 weeks after the last dose of study treatment.
* Participant capable of giving signed informed consent.

Participants with Moderate Hepatic Impairment (Cohort 1):

* Moderate hepatic impairment (of any etiology) and clinically stable for at least 1 month prior to screening.
* Child-Pugh score of 7-9.
* Previous confirmation of liver cirrhosis confirmed by either- Liver biopsy, Imaging technique, or Noninvasive liver assessment consistent with cirrhosis.
* Hepatic impairment needs to be chronic (>6 months), stable.

Matched Healthy Control Participants (Cohort 2):

* Participants will be matched by age plus or minus (±)10 years to a corresponding participant in the hepatic impairment group. Age should remain between 18 and 75 years of age (inclusive).
* Participants will be matched by total body weight ±15 percentage (%) to a corresponding participant in the hepatic impairment group.
* Participants will be matched by gender and race to a corresponding participant in the hepatic impairment group.
* Healthy participant as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and ECG.

Exclusion Criteria:

All Participants:

* Participants are excluded from the study if any of the following medical conditions apply:
* History of cholecystectomy, current symptomatic cholelithiasis or inflammatory gallbladder disease.
* Significant history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history review), clinical laboratory tests, or 12-lead ECG.
* Current clinically significant diarrhea.
* History of gastrointestinal surgery with ileal resection or ileal bypass at any time.
* Any malignancy within the past 5 years except for basal cell or squamous cell carcinoma of the skin disease for 3 years.
* Participants with unstable cardiac function or participants with uncontrolled hypertension.
* Any current medical or psychiatric condition, clinical or laboratory abnormality, or examination finding which may affect study compliance or investigational procedures or possible consequences of the study.
* Administration of any other Ileal bile acid transport (IBAT) inhibitor (including linerixibat) in the 3 months prior to screening.
* For healthy participants, past or intended use of over the counter or prescription medication, including vitamins and dietary or herbal supplements) within 7 days prior to the first dose of study medication.
* Current enrolment in a clinical trial or recent participation in a clinical trial and has received an investigational product within the following time-period prior to study drug administration in the current study: 30 days.
* Positive pregnancy test at screening or at Day -1 in women of childbearing potential.
* Positive human immunodeficiency virus (HIV) antibody test.
* Healthy control participant has corrected interval using the Fridericia's QT correction formula (QTcF) >450 millisecond (msec); or participant with hepatic impairment has a baseline QTcF >480 msec on ECG.
* Regular use of known drugs of abuse or history of drug abuse or dependence within 6 months of the study.
* Moderate (or greater) alcohol consumption defined as one standard drink per day for women and two drinks per day for men.
* History of regular use of tobacco or nicotine-containing products.
* Positive drug/alcohol screen at Screening or at Day -1.
* Where participation in the study would result in donation of blood or blood products more than 500 milliliter (mL) within a 56-day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that contraindicates participation in the study.

Participants with Hepatic Impairment (Cohort 1):

* History of gastric or oesophageal variceal bleeding within the past 6 months and for which varices have not been adequately treated medically or endoscopically.
* Grade 3 ascites (large ascites with marked abdominal distension) refractory to medical therapy.
* Refractory hepatic encephalopathy as judged by the investigator.
* Child-Pugh score of 10 or higher or Child-Pugh score of 6 or lower.
* Hepatopulmonary or hepatorenal syndrome and history of liver transplantation.
* Evidence of active infection, including spontaneous bacterial peritonitis.
* Confirmed hepatocellular carcinoma (HCC) or biliary cancer.
* Alanine amino transferase (ALT) value >3 x upper limit of normal (ULN).
* Platelet count less than (<) 50,000/microliter (μl).

Matched Healthy control participants (Cohort 2):

* Current or chronic history of liver disease or known hepatic or biliary abnormalities and/or confirmed hepatocellular carcinoma or biliary cancer.
* Screening ALT or aspartate aminotransferase (AST) above the upper limit of normal (ULN).
* Elevated bilirubin above the ULN unless this is due to underlying Gilbert's syndrome.
* Presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Plasma area under the concentration-time curve from time zero (pre-dose) to the time of the last quantifiable concentration [AUC(0-t)] following a single dose of linerixibat | Up to Day 3
Maximum observed concentration (Cmax) following a single dose of linerixibat | Up to Day 3

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 14
  AEs and SAEs will be collected
Number of participants with clinically significant change from baseline in electrocardiogram (ECG) | Baseline (Day -1) and up to Day 3
Number of participants with clinically significant change from baseline in vital signs | Baseline (Day -1) and up to Day 3
Number of participants with clinically significant change from baseline in clinical laboratory tests | Baseline (Day -1) and up to Day 3
  Blood samples will be collected for the assessment of clinical laboratory tests
Plasma area under the concentration-time curve from time zero (pre-dose) to 24 hours [AUC (0- 24)] following a single dose of linerixibat | Up to Day 3
Apparent terminal phase half-life (t1/2) of linerixibat | Up to Day 3
Apparent clearance (CL/F) of linerixibat | Up to Day 3
Time to Cmax (tmax) of linerixibat | Up to Day 3
Apparent terminal phase volume of distribution (Vz/F) of linerixibat | Up to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com